CLINICAL TRIAL: NCT05864430
Title: Evaluatıon of The Effıcıency of Sexual and Reproductıve Health Educatıon
Brief Title: Effıcıency of Sexual and Reproductıve Health Educatıon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Nurdan Demirci, PhD RN, Professor, Marmara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MarmaraU-OZ-2023-sexual
Record Dates: First submitted 2023-05-09; First posted 2023-05-18 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Reproductive Health; Sexual Health
Keywords: Sexual Health,; Reproductive Health; Online; DataMatrix; Face-to-face training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Face-to-face Training Group (Experimental): Students in this group will be given face-to-face training on SRH by the principal researcher accompanied by PowerPoint.
  Interventions: Other: Face-to-face Training Group
- DataMatrix supported Face-to-face training group (Experimental): Before starting the training, a QR code including PowerPoint on SRH will be given to the students in the group that receives training with QR code support (on the first slide). Students will be directed to the URL automatically determined by the researcher by scanning the QR code with the camera of their smartphones. Students will follow the lesson with the QR code given simultaneously with the training given during the education process.
  Interventions: Other: DataMatrix supported Face-to-face training group
- Online training group (Experimental): The students in the online training group will be given training on SRH/RES on an online platform accompanied by PowerPoint by the principal researcher.
  Interventions: Other: Online training group

INTERVENTIONS:
Other: Face-to-face Training Group — The training will take approximately 3 hours. The training will be done interactively, allowing students to talk to each other and ask questions, and will end with 10 minutes of time for students' questions.
  Arms: Face-to-face Training Group
Other: DataMatrix supported Face-to-face training group — Students will follow the lesson with the QR code given simultaneously with the training given during the education process. The training will be held in such a way that the students will be given the opportunity to ask questions and will end with 10 minutes of time to be given to the questions of the students.
  Arms: DataMatrix supported Face-to-face training group
Other: Online training group — The training will take approximately 3 hours. The training will be done interactively, allowing students to talk to each other and ask questions, and will end with 10 minutes of time for students' questions.
  Arms: Online training group

SUMMARY:
The youth period is a period when information and education are important. Reproductive and sexual health problems have an important place in aging health problems in youth (Gölbaşlı 2003). All over the world, STIs are most common in the 20-24 age group, followed by the 15-19 and 25-29 age groups. STIs are the most common disease in many countries, especially among young people between the ages of 15-29 (Topbaş et al. 2003). STIs, which are one of the factors that negatively affect public health; are infections transmitted from person to person through sexual contact. According to WHO estimates, approximately 350 million people suffer from curable STIs each year, and the incidence and prevalence of STIs among young people in developed and developing countries are increasing.

Although young adults are generally at risk, STIs are most common in people aged 15-49. They have a very important place in terms of human health because they are frequently seen, difficult to diagnose, and cause serious complications when not treated. Incomplete and incorrect information among people who start sexual intercourse at an early age causes difficulties in the prevention of these diseases (Özalp et al. 2012).

Having sexual intercourse at an early age, being polygamous, having special sexual preferences, being with or having sex with those who have paid for sexual intercourse, and not using condoms are among the risk factors for STIs (Siyez 2009).

We can say that the age period in which STIs are common is parallel to sexual activity. In addition to various socio-demographic factors, it is likely that the most provoking issue in this period is the lack of knowledge of young people (Karaköse and Aydın 2011).

In the STD guide published by the CDC, it is recommended to evaluate the people who constitute the risk group in the prevention of these diseases and to provide education and counseling (CDC, 2020). In this context, training to increase the level of knowledge and awareness of young people, who are one of the high-risk groups in society in terms of STD, is important in terms of reducing risky sexual behaviors, early diagnosis, and treatment.

Based on all these reasons; It is aimed to evaluate the effectiveness of sexual and reproductive health education given to university students.

DETAILED DESCRIPTION:
During the International Conference on Population and Development held in Cairo in 1994, SRH was covered extensively for the first time and the scope of reproductive and sexual health was expanded (ICPD, 1994). If the concepts that make up the SRH of adolescents and young people are examined, the term sexual health is used to describe the absence of disease and disability related to sexuality and the sense of sexual well-being. It has been defined as a positive combination of the physical, emotional, intellectual, and social aspects of sexuality. Sexuality influences thoughts, feelings, interactions, and actions between individuals, motivating people to find love, contact, warmth, and intimacy. Sexuality can be expressed in many different ways and it has been determined that it is closely linked to the environment in which people live.

Reproductive health is defined as a state of complete physical, mental and social well-being and not merely the absence of disease or infirmity in all matters related to the reproductive system, its functions and processes. Reproductive health therefore means that people can live a satisfying and safe sex life and have the freedom to decide when and how often to use their reproductive capacity. Men and women have the right to have access to safe, effective, affordable and acceptable methods of family planning, the right to be informed, and the right to access health services that will ensure a safe pregnancy and delivery, and the chance to have a healthy baby.

The scope of reproductive health includes methods, techniques and services that contribute to reproductive health and welfare by providing reproductive health care, preventing and solving reproductive health problems. The aim of reproductive health includes not only reproductive and STI-related counseling and care, but also sexual health, which is to improve life and personal relationships (WHO, 2006).Adolescents and young people, like all individuals, have the right to make decisions concerning their own bodies and to access services that support this right. Ensuring sexual and reproductive health for all depends on the realization of sexual and reproductive rights based on human rights (Engel et al., 2019).

Based on all these reasons; In this study, it is aimed to evaluate the effectiveness of sexual and reproductive health education given to university students.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the research,
* Have not taken Sexual Health, Infectious Diseases course before
* Students without communication barriers will be included.

Exclusion Criteria:

* Incorrect or incomplete form filling
* The participant's wish to withdraw from the study

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 165 (Actual)
Dates: Start 2022-05-15 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Participant Identification Form Diagnostic Form | 5 Months
  The participant identification form, which includes the introductory characteristics of the students, was prepared by the researchers in line with the literature (Altay et al., 2020; Vongxay et al., 2019). The form includes students' socio-demographic characteristics, their status of obtaining information about SRH and sources of information, their experiences with SRH and their thoughts on sexual intercourse. The form consists of 28 questions in total.

SECONDARY OUTCOMES:
Sexual Health Knowledge Test | 5 Months
  It was developed by Petili and Gölbaşı in 2017, and its validity-reliability has been made. The test consists of 40 multiple-choice questions and includes 12 sub-dimensions.

OTHER OUTCOMES:
Reproductive Health Scale for Turkish Adolescents | 5 Months
  It was developed by Saydam et al. in 2010 to measure the reproductive behavior of adolescents in a valid and reliable way. SRQ consists of six sub-dimensions and a total of 34 items. Scale sub-dimensions; Partner Selection, Values in Developing Protective Behavior, Communication with a Sexual Spouse (Partner), Counseling, Trust and Protection from Sexually Transmitted Diseases.

CONTACTS AND LOCATIONS:
Overall Officials: Tuğba Öz, Principal Investigator — ev
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Package of Sexual and Reproductive Health and Rights Interventions-What Does It Mean for Adolescents? — https://europepmc.org/article/med/31761003
- See also: What do we know about sexting, and when did we know it? — https://pubmed.ncbi.nlm.nih.gov/31648755/